CLINICAL TRIAL: NCT02312258
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind Study of Oral Ixazomib Maintenance Therapy After Initial Therapy in Patients With Newly Diagnosed Multiple Myeloma Not Treated With Stem Cell Transplantation
Brief Title: A Study of Oral Ixazomib Maintenance Therapy in Participants With Newly Diagnosed Multiple Myeloma (NDMM) Not Treated With Stem Cell Transplantation (SCT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C16021; U1111-1160-1702 (Registry Identifier: WHO); 2014-001394-13 (EudraCT Number); REec-2015-1414 (Registry Identifier: REec); JapicCTI-152873 (Registry Identifier: JapicCTI); 153300410A0048 (Registry Identifier: RNEC); 1046003327 (Registry Identifier: TCTIN); SNCTP000001745 (Registry Identifier: SNCTP); 15/NE/0167 (Registry Identifier: NRES); 182602 (Registry Identifier: HC-CTD)
Record Dates: First submitted 2014-12-05; First posted 2014-12-09 (Estimated); Results first posted 2020-11-10 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Multiple Myeloma
Keywords: Drug Therapy
MeSH Terms: conditions — Multiple Myeloma | interventions — ixazomib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Ixazomib placebo-matching capsule, orally, once on Days 1, 8, and 15 of each 28-day cycle from Cycles 1 through 26.
  Interventions: Drug: Placebo
- Ixazomib (Experimental): Ixazomib 3 mg, capsule, orally, once on Days 1, 8, and 15 of each 28-day cycle from Cycles 1 to 4 that may have been escalated to 4 mg thereafter up to Cycle 26.
  Interventions: Drug: Ixazomib

INTERVENTIONS:
Drug: Placebo — Ixazomib placebo-matching capsules.
  Arms: Placebo
Drug: Ixazomib — Ixazomib capsules.
  Arms: Ixazomib

SUMMARY:
The purpose of this study is to determine the effect of ixazomib maintenance therapy on progression free survival (PFS) compared with placebo, in participants with NDMM who have had a major response (complete response [CR], very good partial response [VGPR], or partial response [PR]) to initial therapy and who have not undergone SCT.

DETAILED DESCRIPTION:
The drug being tested in this study is called ixazomib citrate. Ixazomib citrate is being tested to slow progressive disease (PD) and improve overall survival in people who have NDMM who have had a major positive response to initial therapy and have not undergone SCT. This study will look at the effect of ixazomib citrate has on the length of time that participants are free of PD and their overall survival.

The study will enrol approximately 700 participants. Participants will be randomly assigned (by chance, like flipping a coin) in 3:2 ratio to Ixazomib or matching placebo groups-which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* Ixazomib citrate initiates at 3 mg which will be escalated to 4 mg with cycle 5 day 1
* Placebo (dummy inactive pill) - this is a capsule that looks like the study drug but has no active ingredient

All participants will be asked to take one capsule on Days 1, 8 and 15 of each 28-day cycle. The treatment period will be approximately 24 months (equivalent to 26 cycles) or until patients experience PD or unacceptable toxicities, whichever occurs first.

This multi-center trial will be conducted worldwide. The overall time to participate in this study is approximately 78 to 106 months. Participants will make 28 visits to the clinic during the treatment period and will continue to make follow-up visits every 4 weeks until the next line of therapy begins. Participants will also be contacted by telephone every 12 weeks after last treatment visit for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Adult male or female participants 18 years or older with a confirmed diagnosis of symptomatic newly diagnosed multiple myeloma (NDMM) according to standard criteria.
2. Completed 6 to 12 months (± 2 weeks) of initial therapy, during which the participant was treated to best response, defined as the best response maintained for 2 cycles after the M-protein nadir is reached.
3. Documented major response (PR, VGPR, CR) according to the International Myeloma Working Group (IMWG) uniform response criteria, version 2011, after this initial therapy.
4. Female participants who:

   * Are postmenopausal for at least 1 year before the screening visit, OR
   * Are surgically sterile, OR
   * If they are of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [eg, calendar, ovulation, symptothermal, postovulation methods] and withdrawal are not acceptable methods of contraception.)

   Male participants, even if surgically sterilized (that is, status postvasectomy), who:
   * Agree to practice effective barrier contraception during the entire study Treatment period and through 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence, when this is in line with the preferred and usual lifestyle of the participant. (Periodic abstinence [example, calendar, ovulation, symptothermal, postovulation methods for the female partner] and withdrawal are not acceptable methods of contraception.)
5. Voluntary written consent must be given before performance of any study-related procedure not part of standard medical care, with the understanding that consent may be withdrawn by the participant at any time without prejudice to future medical care.
6. Complete documentation of the details of the initial therapy before randomization including cytogenetics and International Staging System (ISS) is available.
7. Eastern Cooperative Oncology Group Performance Status of 0 to 2.
8. Suitable venous access for the study-required blood sampling and consent for the specific amounts that will be taken.
9. Is willing and able to adhere to the study visit schedule and other protocol requirements including blood sampling and bone marrow aspiration.
10. Must meet the following clinical laboratory criteria at study entry:

    * Absolute neutrophil count (ANC) greater than or equal to (≥) 1,000 per cubic millimeter (/mm^3) without growth factor support and platelet count ≥75,000/mm^3. Platelet transfusions to help participants meet eligibility criteria are not allowed within 3 days before randomization.
    * Total bilirubin less than or equal to (≤) 1.5*the upper limit of the normal range (ULN).
    * Alanine aminotransferase and aspartate aminotransferase ≤ 3*ULN.
    * Calculated creatinine clearance ≥ 30 milliliter per minute (mL/min) (using the Cockcroft-Gault equation).

Exclusion Criteria:

1. Multiple myeloma that has relapsed after, or was not responsive to, initial therapy.
2. Prior SCT.
3. Radiotherapy within 14 days before randomization.
4. Diagnosed or treated for another malignancy within 5 years before randomization or previous diagnosis with another malignancy. Participants with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
5. Female participants who are lactating and breastfeeding or have a positive serum pregnancy test during the Screening period.
6. Major surgery within 14 days before randomization.
7. Central nervous system involvement.
8. Infection requiring intravenous (IV) antibiotic therapy or other serious infection within 14 days before randomization.
9. Diagnosis of Waldenstrom's macroglobulinemia, polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes syndrome (POEMS), plasma cell leukemia, primary amyloidosis, myelodysplastic syndrome, or myeloproliferative syndrome.
10. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, uncontrolled congestive heart failure, unstable angina, or myocardial infarction within the past 6 months.
11. Systemic treatment with strong cytochrome P450 3A (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital) or St. John's wort within 14 days before randomization.
12. Ongoing or active infection, known human immunodeficiency virus (HIV) positive, active hepatitis B or C infection.
13. Comorbid systemic illnesses or other severe concurrent disease that, in the judgment of the investigator, would make the participant inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens (example, PN that is Grade 1 with pain or Grade 2 or higher of any cause).
14. Psychiatric illness or social situation that would limit compliance with study requirements.
15. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent.
16. Inability to swallow oral medication, inability or unwillingness to comply with the drug administration requirements, or gastrointestinal (GI) procedure that could interfere with the oral absorption or tolerance of treatment.
17. Treatment with any investigational products within 30 days before randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 706 (Actual)
Dates: Start 2015-04-09 (Actual); Primary Completion 2019-08-12 (Actual); Study Completion 2022-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (275):
- United States (23):
  - Robert A Moss MD FACP Inc, Fountain Valley, California
  - UCLA Medical Hematology and Oncology, Los Angeles, California
  - North County Oncology Medical Clinic Inc, Oceanside, California
  - Ventura County Hematology Oncology Specialists, Oxnard, California
  - Emad Ibrahim, MD, Inc, Redlands, California
  - Global Cancer Research Institute (GCRI), Inc., San Jose, California
  - Central Coast Medical Oncology Corporation, Santa Maria, California
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Siouxland Hematology - Oncology Associates LLP, Sioux City, Iowa
  - Appalachian Regional Healthcare, Hazard, Kentucky
  - New England Cancer Specialists, Scarborough, Maine
  - Saint Agnes Hospital - Baltimore - Hunt - PPDS, Baltimore, Maryland
  - University Hospital of Wales -, Bethesda, Maryland
  - Tufts Medical Center - PPDS, Boston, Massachusetts
  - Herbert-Herman Cancer Center, Lansing, Michigan
  - Clinical Research Alliance Inc, New York, New York
  - New York Presbyterian Hospital - Weill-Cornell, New York, New York
  - Cancer Care of WNC PA, Asheville, North Carolina
  - UPMC Cancer Pavillion, Pittsburgh, Pennsylvania
  - HOPE Cancer Center of East Texas, Tyler, Texas
  - Swedish Cancer Institute, Seattle, Washington
  - W VA University Mary Babb Randolph Cancer Center, Morgantown, West Virginia
- Argentina (5):
  - Hospital Universitario Austral, Buenos Aires, Ciudad Autonoma de BuenosAires
  - Hospital Italiano de Buenos Aires, Buenos Aires, Ciudad Autonoma de BuenosAires
  - Centro de Educacion Medica e Investigaciones Clinicas "Norberto Quirno" (CEMIC), Buenos Aires, Ciudad Autonoma de BuenosAires
  - Sanatorio Allende S.A., Córdoba
  - Hospital Iturraspe, Santa Fe
- Australia (3):
  - St Vincents Hospital Melbourne - PPDS, Fitzroy, Victoria
  - Frankston Hospital, Frankston, Victoria
  - The Alfred Hospital, Melbourne, Victoria
- Austria (4):
  - Universitatsklinikum Innsbruck, Innsbruck, Tyrol
  - Paracelsus Medizinische Privatuniversitat, Salzburg
  - Medizinische Universitat Wien (Medical University of Vienna), Vienna
  - Klinikum Wels-Grieskirchen GmbH, Wels
- Belgium (3):
  - Universitair Ziekenhuis Brussel - PIN, Brussels, Brussels Capital
  - UZ Brussel, Brussels, Brussels Capital
  - Cliniques Universitaires Saint-Luc, Brussels, Brussels Capital
- Brazil (28):
  - Del-pesti Centrumkorhaz- Orszagos Hematologiai és Infektologiai Intezet, Salvador, Estado de Bahia
  - Hospital Das Clinicas Da Universidade Federal de Goias, Goiânia, Goiás
  - Hospital Das Clinicas Da UFMG, Belo Horizonte, Minas Gerais
  - Liga Paranaense de Combate Ao Cancer - Hospital Erasto Gaertner, Curitiba, Paraná
  - Liga Norte Riograndense Contra O Cancer, Natal, Rio Grande do Norte
  - Universidade de Caxias do Sul, Caxias do Sul, Rio Grande do Sul
  - Associacao Hospital de Caridade Ijui, Ijuí, Rio Grande do Sul
  - American Oncology Partners of Maryland, PA, Passo Fundo, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre (HCPA) - PPDS, Porto Alegre, Rio Grande do Sul
  - Mae de Deus Center Hospital Giovanni Battista, Porto Alegre, Rio Grande do Sul
  - Hospital Sao Lucas Da Pontificia Universidade Catolica Do Rio Grande Do Sul (PUCRS), Porto Alegre, Rio Grande do Sul
  - Instituto Joinvilense de Hematologia E Oncologia, Joinville, Santa Catarina
  - Fundacao PIO XII, Barretos, São Paulo
  - Universidade Estadual de Campinas, Campinas, São Paulo
  - Hospital Amaral Carvalho, Jaú, São Paulo
  - Faculdade de Medicina Do ABC, Santo André, São Paulo
  - HEMORIO - Unidade de Pesquisa Clinica, Rio de Janeiro
  - Instituto Nacional de Cancer, Rio de Janeiro
  - Fundação Antônio Prudente - AC Camargo Câncer Center, Rio de Janeiro
  - Hospital de Base Da Faculdade de Medicina de Sao Jose Do Rio Preto, São José do Rio Preto
  - Instituto de Ensino E Pesquisa Sao Lucas, São Paulo
  - Hospital Sirio Libanes, São Paulo
  - Ealing Hospital, São Paulo
  - Clinica Sao Germano, São Paulo
  - Hospital das Clinicas da Faculdade de Medicina da Universidade de Sao Paulo, São Paulo
  - Hospital Israelita Albert Einstein, São Paulo
  - Hospital Santa Marcelina, São Paulo
- Canada (4):
  - Royal Victoria Regional Health Centre, Barrie, Ontario
  - William Osler Health Centre, Brampton, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - McGill University Health Center, Montreal, Quebec
- Chile (4):
  - Hospital Amaral Carvalho, Temuco, Región de la Araucanía
  - Instituto Nacional Del Cancer, Santiago
  - Centro Internacional de Estudios Clinicos, Santiago
  - Centro de Investigaciones Clinicas Vina del Mar, Viña del Mar
- China (12):
  - Hospital de Clinicas de Passo Fundo, Nanjing, Jiangsu
  - Ruijin Hospital Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou, Zhejiang
  - Beijing Chaoyang Hospital Capital Medical University, Beijing
  - Peking University Third Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The First Affiliated Hospital, College of Medicine, Zhejiang University, Hangzhou
  - Renji Hospital Shanghai Jiaotong University School of Medicine, Shanghai
  - Shanghai Chang Zheng Hospital, Shanghai
  - Hospital São Rafael, Shenyang
  - Second Hospital of Shanxi Medical University, Taiyuan
  - James Lind Centro de Investigación del Cáncer, Wuhan
- Colombia (3):
  - Hospital Pablo Tobon Uribe, Medellín, Antioquia
  - Hospital Universitario San Ignacio, Bogotá, Bogota D.C.
  - Instituto Nacional de Cancerologia Colombia, Bogota, Cundinamarca
- Croatia (3):
  - Clinical Hospital Dubrava, Zagreb, City of Zagreb
  - Clinical Hospital Center Rijeka, Rijeka
  - Clinical Hospital Center Zagreb - PPDS, Zagreb
- Czechia (6):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové, Kralovehradeck Kraj
  - Fakultni nemocnice Kralovske Vinohrady, Prague, Praha, Hlavni Mesto
  - Fakultni nemocnice Brno, Brno
  - Fakultni nemocnice Olomouc, Olomouc
  - Fakultni nemocnice Ostrava, Ostrava
  - Vseobecna fakultni nemocnice v Praze, Prague
- Denmark (4):
  - Jiangsu Province Hospital (the First Affiliated Hospital With Nanjing Medical University), Copenhagen, Capital
  - Aarhus Universitetshospital Århus Sygehus, Aarhus N
  - Regionshospitalet Holstebro, Holstebro
  - Odense Universitetshospital, Odense
- France (11):
  - Hopital Antoine Beclere, Clamart, Hauts-de-Seine
  - Hotel Dieu, Nantes, Loire-Atlantique
  - CHRU Nancy, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - CHRU Dijon Complexe Du Bocage, Dijon
  - Hopital Saint Vincent de Paul GHICL, Lille
  - CHRU Lille, Lille
  - Hopital de la Pitie Salpetriere, Paris
  - Groupe Hospitalier Necker Enfants Malades, Paris
  - Hopital Haut Leveque, Pessac
  - Hopital Jean Bernard, Poitiers
  - CHRU Rennes, Rennes
- Germany (17):
  - Universitatsklinikum Ulm, Ulm, Baden-Wurttemberg
  - Schwarzwald Baar Klinkum Villingen-Schwenningen GmbH, Villingen-Schwenningen, Baden-Wurttemberg
  - Hamatologische Onkologische Gemeinschaftspraxis Dr. Brudler, Dr. Heinrich, Dr. Bangerter, Augsburg, Bavaria
  - Internistisch Hamatologische und Internistische Praxis, Herrsching am Ammersee, Bavaria
  - LMU Klinikum der Universitat Munchen, München, Bavaria
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Universitatsklinikum Essen, Essen, North Rhine-Westphalia
  - Gemeinschaftspraxis fur Hamatologie und Onkologie, Münster, North Rhine-Westphalia
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz, Mainz, Rhineland-Palatinate
  - Universitat Des Saarlandes, Homburg, Saarland
  - Onkologie Aschaffenburg, Aschaffenburg
  - Charite - Universitatsmedizin Berlin, Berlin
  - Medizinisches Versorgungszentrum Onkologischer Schwerpunkt, Berlin
  - Klinikum Landshut, Landshut
  - Klinikum rechts der Isar der Technischen Universitat Munchen, München
  - Praxis Pihusch Medizinisches Versorgungszentrum GbR, Rosenheim
  - Gemeinschaftspraxis Dr. med. R. Schlag & Dr. med. B. Schottker & Dr. med. J. Haas, Würzburg
- Greece (6):
  - University of Athens Medical School - Regional General Hospital Alexandra, Athens, Attica
  - Evangelismos General Hospital of Athens, Athens
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Larissa, Larissa
  - Theageneio Anticancer Oncology Hospital of Thessaloniki, Thessaloniki
  - Georgios Papanikolaou General Hospital of Thessaloniki, Thessaloniki
- Hungary (4):
  - Semmelweis Egyetem, Budapest
  - Klinika Hematologii, Szpital Uniwersytecki Nr 2 im. Jana Biziela w Bydgoszczy, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Szegedi Tudomanyegyetem Szent-Gyorgyi Albert Klinikai Kozpont, Szeged
- Israel (10):
  - Rigshospitalet, Beer Yaakov
  - Shamir Medical Center Assaf Harofeh, Beersheba
  - Bnai Zion Medical Center, Haifa
  - Hadassah Medical Center - PPDS, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center - PPDS, Petah Tikva
  - Chaim Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Tel Aviv
  - Assuta Medical Centers, Tel Aviv
  - Baruch Padeh Poriya Medical Center, Tiberias
- Italy (15):
  - Ospedale Casa Sollievo Della Sofferenza IRCCS, San Giovanni Rotondo, Apulia
  - AORN A Cardarelli, Napoli, Campania
  - Azienda Ospedaliero Universitaria Di Bologna - Policlinico S Orsola Malpighi, Bologna, Emilia-Romagna
  - Ospedale Infermi di Rimini, Rimini, Emilia-Romagna
  - IRCCS Az. Osp. Universitaria San Martino- IST, Genoa, Liguria
  - ASST degli Spedali Civili di Brescia - Spedali Civili di Brescia - INCIPIT - PIN, Brescia, Lombardy
  - ASST Grande Ospedale Metropolitano Niguarda - Presidio Ospedaliero Ospedale Niguarda Ca' Granda, Milan, Lombardy
  - Azienda Ospedaliero Universitaria Policlinico Vittorio Emanuele, Catania, Sicily
  - Azienda Ospedaliero Universitaria Pisana, Pisa, Tuscany
  - Azienda Ospedaliera S Maria Di Terni, Terni, Umbria
  - Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona-Umberto I G.M. Lancisi G. Salesi, Ancona
  - Azienda Ospedaliera Universitaria Careggi, Florence
  - Azienda Ospedaliero Universitaria di Parma, Parma
  - Ospedale Santa Maria Delle Croci, Ravenna
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Japan (20):
  - Ogaki Municipal Hospital, Ōgaki, Gihu
  - Kobe City Medical Center General Hospital, Kobe, Hyōgo
  - Hitachi General Hospital, Hitachi, Ibaraki
  - Nara Hospital Kinki University Faculty of Medicine, Ikoma, Nara
  - National Hospital Organization Okayama Medical Center, Okayama, Okayama-ken
  - Juntendo University Hospital, Bunkyo, Tokyo
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo
  - National Hospital Organization Kyushu Medical Center, Fukuoka
  - Fukushima Medical University Hospital, Fukushima
  - National Hospital Organization Mito Medical Center, Ibaraki
  - Kurume University Hospital, Kurume
  - Shizuoka Cancer Center, Nagaizumi-chō
  - Japanese Red Cross Nagoya Daiichi Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Japanese Red Cross Narita Hospital, Narita-shi
  - Niigata Cancer Center Hospital, Niigata
  - Osaka Saiseikai Nakatsu Hospital, Osaka
  - National Hospital Organization Disaster Medical Center, Tachikawa
  - Toyohashi Municipal Hospital, Toyohashi
  - Yamanashi Prefectural Central Hospital, Yamanashi
- Mexico (5):
  - Centro de Investigacion Farmaceutica Especializada de Occidente, SC - PPDS, Guadalajara, Jalisco
  - Hospital Y Clinica OCA Sociedad Anonima de Capital Variable, Monterrey, Nuevo León
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City
  - Oaxaca Site management Organization (OSMO) - PPDS, Oaxaca City
- Poland (4):
  - Shengjing Hospital of China Medical University, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - MTZ Clinical Research Sp z o o - PRATIA - PPDS, Warsaw, Masovian Voivodeship
  - Samodzielny Publiczny Zaklad Opieki Zdrowotnej Zespol Szpitali Miejskich, Chorzów
  - Samodzielny Publiczny Szpital Kliniczny Nr 1 we Wroclawiu, Wroclaw
- Portugal (7):
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil, E.P.E., Lisbon, Lisbon District
  - Hospital Garcia de Orta, Almada
  - Hospital de Braga, Braga
  - Champalimaud Cancer Center, Lisbon
  - Centro Hospitalar do Porto - Hospital de Santo Antonio, Porto
  - Instituto Portugues de Oncologia Do Porto Francisco Gentil Epe - PPDS, Porto
  - Centro Hospitalar de Sao Joao EPE, Porto
- Russia (5):
  - State Medical and Preventive Treatment Institution Kirov Regional Clinical Oncology Dispensary, Kirov
  - Stavropol Regional Clinical Oncology Centre Pyatigorsk Affiliate, Pyatigorsk
  - Ryazan Regional Clinical Hospital, Ryazan
  - Russian Research Institute of Hematology and Blood Transfusion, Saint Petersburg
  - City Center of MS Treatment based on Saint-Petersburg City Clinical Hospital #31, Saint Petersburg
- Serbia (4):
  - Tongji Hospital Tongji Medical College Huazhong University of Science and Technology, Belgrade
  - Clinical Hospital Center ''Bezanijska Kosa'', Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Soroka University Medical Centre, Niš
- Singapore (2):
  - National University Hospital, Singapore
  - Singapore General Hospital (SGH), Singapore
- South Africa (3):
  - Medical Oncology Centre of Rosebank, Johannesburg, Gauteng
  - Albert Alberts Stem Cell Transplant Centre, Pretoria, Gauteng
  - Mary Potter Oncology Centre, Pretoria, Gauteng
- South Korea (6):
  - National Cancer Center, Goyang-si, Gyeonggido
  - Gachon University Gil Medical Center, Incheon
  - Seoul National University Hospital, Seoul
  - Severance Hospital Yonsei University Health System - PPDS, Seoul
  - Samsung Medical Center - PPDS, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (13):
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Quironsalud Madrid, Pozuelo de Alarcón, Madrid, Communidad Delaware
  - Clinica Universidad Navarra, Pamplona, Navarre
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario de La Princesa, Madrid
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario HM Sanchinarro CIOCC, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Complejo Asistencial Universitario de Salamanca H. Clinico, Salamanca
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- Sweden (4):
  - Karolinska Universitetssjukhuset Huddinge, Stockholm, Södermanland County
  - Karolinska Universitetssjukhuset Solna, Stockholm, Södermanland County
  - Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County
  - Skanes Universitetssjukhus Lund, Lund
- Spital STS AG, Thun, Switzerland
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- Thailand (3):
  - Ramathibodi Hospital, Bangkok, Bangkok
  - Chulalongkorn University, Bangkok
  - Maharaj Nakorn Chiang Mai Chiang Mai University, Chiang Mai
- Turkey (Türkiye) (4):
  - Hacettepe Universitesi Tip Fakultesi Hastanesi, Ankara
  - Ankara University Medical Faculty PPDS, Ankara
  - Istanbul Universitesi Istanbul Tip Fakultesi Hastanesi, Istanbul
  - Dokuz Eylul University Medical Faculty, Izmir
- United Kingdom (26):
  - Belfast City Hospital, Belfast, Antrim
  - Birmingham Heartlands Hospital, West Malling, Birmingham
  - Bristol Haematology and Oncology Centre, Bristol, Bristol, City of
  - Royal Bournemouth Hospital, Bournemouth, Dorset
  - Queen Alexandra Hospital, Portsmouth, Hampshire
  - Kent and Canterbury Hospital, Canterbury, Kent
  - Barts Health NHS Trust, London, London, City of
  - University College London, London, London, City of
  - Kings College Hospital, London, London, City of
  - Hammersmith Hospital, London, London, City of
  - Hillingdon Hospital, Uxbridge, London, City of
  - Churchill Hospital, Oxford, Oxfordshire
  - New Cross Hospital, Wolverhampton, Staffordshire
  - Royal Marsden Hospital - Surrey, Sutton, Surrey
  - Royal United Hospital, Bath
  - Ulster Hospital, Belfast
  - Southmead Hospital, Bristol
  - University Clinical Center Nis, Cardiff
  - West Middlesex University Hospital, Isleworth
  - Leicester Royal Infirmary, Leicester
  - Chelsea and Westminster NHS Trust, London
  - Manchester Royal Infirmary - PPDS, Manchester
  - Northwick Park Hospital, Middlesex
  - The Royal Oldham Hospital - PPDS, Oldham
  - University Clinical Center of Serbia - PPDS, Southall
  - Singleton Hospital - PPDS, Swansea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Paiva B, Manrique I, Dimopoulos MA, Gay F, Min CK, Zweegman S, Spicka I, Teipel R, Mateos MV, Giuliani N, Cavo M, Hopkins CR, Fu W, Suryanarayan K, Vorog A, Li C, Wang B, Estevam J, Labotka R, Dash AB. MRD dynamics during maintenance for improved prognostication of 1280 patients with myeloma in the TOURMALINE-MM3 and -MM4 trials. Blood. 2023 Feb 9;141(6):579-591. doi: 10.1182/blood.2022016782. PMID 36130300
- [Derived] Dimopoulos MA, Spicka I, Quach H, Oriol A, Hajek R, Garg M, Beksac M, Bringhen S, Katodritou E, Chng WJ, Leleu X, Iida S, Mateos MV, Morgan G, Vorog A, Labotka R, Wang B, Palumbo A, Lonial S; TOURMALINE-MM4 study group. Ixazomib as Postinduction Maintenance for Patients With Newly Diagnosed Multiple Myeloma Not Undergoing Autologous Stem Cell Transplantation: The Phase III TOURMALINE-MM4 Trial. J Clin Oncol. 2020 Dec 1;38(34):4030-4041. doi: 10.1200/JCO.20.02060. Epub 2020 Oct 6. PMID 33021870

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study from 09 April 2015 to 26 August 2022.
Pre-assignment Details: Participants with newly diagnosed multiple myeloma not treated with stem cell transplantation (SCT) were enrolled and randomized in a 3:2 ratio to receive ixazomib or placebo respectively.
Period: Overall Study
Arm/Group | Placebo | Ixazomib
Started | 281 | 425
Safety Population (The safety population was defined as all participants who received at least 1 dose of ixazomib or placebo. Three placebo participants who erroneously received a single dose of ixazomib were included in the ixazomib arm of the safety population.) | 276 | 426
Completed | 0 | 0
Not Completed | 281 | 425
Not completed — Lost to Follow-up | 8 | 8
Not completed — Withdrawal by Patient | 49 | 76
Not completed — Reason not Specified | 107 | 159
Not completed — Missing | 2 | 1
Not completed — Death | 115 | 181

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population included all participants who were randomized and had post-randomization data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ixazomib | Total
Number analyzed (Participants) | 281 | 425 | 706
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.8 (6.77) | 72.3 (6.87) | 72.5 (6.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 126 | 203 | 329
  Male | 155 | 222 | 377
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 36 | 46 | 82
  Not Hispanic or Latino | 237 | 366 | 603
  Unknown or Not Reported | 8 | 13 | 21
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 39 | 63 | 102
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 5 | 15 | 20
  White | 227 | 330 | 557
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 9 | 15 | 24
Region of Enrollment [Count of Participants; unit: Participants]
  Australia | 11 | 9 | 20
  China | 3 | 6 | 9
  Japan | 15 | 17 | 32
  Singapore | 4 | 8 | 12
  Korea, Republic Of | 10 | 17 | 27
  Taiwan, Province Of China | 3 | 5 | 8
  Thailand | 2 | 8 | 10
  Austria | 2 | 3 | 5
  Belgium | 0 | 1 | 1
  Czech Republic | 31 | 38 | 69
  Denmark | 1 | 5 | 6
  France | 10 | 6 | 16
  Germany | 5 | 6 | 11
  Greece | 50 | 63 | 113
  Hungary | 5 | 7 | 12
  Israel | 5 | 11 | 16
  Italy | 18 | 34 | 52
  Poland | 2 | 13 | 15
  Portugal | 6 | 10 | 16
  Russia | 2 | 6 | 8
  Serbia | 11 | 13 | 24
  South Africa | 2 | 5 | 7
  Spain | 23 | 25 | 48
  Sweden | 3 | 3 | 6
  Switzerland | 1 | 1 | 2
  Turkey | 4 | 8 | 12
  United Kingdom | 20 | 46 | 66
  Argentina | 2 | 2 | 4
  Brazil | 16 | 27 | 43
  Chile | 4 | 7 | 11
  Colombia | 1 | 2 | 3
  Canada | 4 | 3 | 7
  Mexico | 2 | 4 | 6
  United States | 3 | 6 | 9

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time from the date of randomization to the date of first documentation of progressive disease (PD) or death from any cause, as evaluated by an independent review committee (IRC) according to International Myeloma Working Group (IMWG) criteria, or death due to any cause, whichever occurs first. Per IMWG criteria, PD is defined as, increase of 25% of lowest response value in one or more of following criteria: serum M-component (absolute increase ≥0.5 g/ deciliter (dL)); or urine M-component (absolute increase ≥200 mg/24-hour); difference between involved and uninvolved free light chains (FLC) levels (absolute increase >10 mg/dL); or bone marrow plasma cell percentage (absolute plasma cell percentage ≥10%); development of new/ increase in size of existing bone lesions or soft tissue plasmacytoma; or development of hypercalcemia (corrected serum calcium >11.5mg/dL).
Time Frame: From randomization until PD or death (up to 52 months)
Population: ITT Population included all participants who were randomized and had post-randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 281 | 425
months | 9.4 [8.51 to 11.47] | 17.4 [14.78 to 20.30]

2. Secondary Outcome: Overall Survival (OS)
Description: OS was measured as the time from the date of randomization to the date of death.
Time Frame: From the date of randomization and every 12 weeks after PD on next-line therapy until death (up to 88 months)
Population: ITT Population included all participants who were randomized and had post-randomization data.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Placebo: Ixazomib 3 mg, capsule, orally, once on Days 1, 8, and 15 of each 28-day cycle from Cycles 1 through 26.
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 281 | 425
months | 69.5 [56.67 to 75.17] | 64.8 [54.87 to 74.84]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib; Test type: Superiority; p = 0.473, Log Rank; Hazard Ratio (HR) = 1.090, 95% CI 2-sided [0.861 to 1.381]; P-value comparing OS between treatment groups was based on log-rank test stratified by initial therapy (proteasome inhibitor-containing or not), International Staging System (ISS) stage before initial therapy (stage I or II vs stage III), age (<75 versus [vs] >=75 years) at randomization, and best response to initial therapy (complete response (CR) or very good partial response (VGPR) vs partial response (PR)). Hazard ratio was based on an unadjusted Cox's proportional hazard regression model stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 versus[vs] >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR), comparing the hazard rate of ixazomib arm over the hazard rate of placebo arm. A less than 1 hazard ratio was to be considered statistically significant

3. Secondary Outcome: Percentage of Participants Who Achieve or Maintain Any Best Response Category During the Treatment Period
Description: Response was assessed according to IMWG criteria based on IRC assessment. Best response included PR, VGPR and CR. PR= >=50% reduction of serum M protein and >=90% or <200 mg reduction urinary M protein in 24-hour, or >50% decrease in difference between involved and uninvolved FLC levels, or >50% reduction in bone marrow plasma cells, if bone marrow plasma cells >30% and >50% reduction in size of soft tissue plasmacytomas at baseline. VGPR= >90% reduction (<100 mg/24-hour) in serum M-protein + urine M-protein detectable by immunofixation but not on electrophoresis. Complete response= >5% plasma cells in myelogram with absence of paraprotein in serum and urine according to immunofixation.
Time Frame: Up to 27 months
Population: ITT Population included all participants who were randomized and had post-randomization data. The percentages are rounded off to the single nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 281 | 425
percentage of participants
  PR | 29 | 25
  VGPR | 37 | 34
  CR | 28 | 31

4. Secondary Outcome: Time to Progression (TTP)
Description: TTP is defined as the time from the date of randomization to the date of first documentation of PD, using IMWG criteria.
Time Frame: From randomization until PD or death (up to 52 months)
Population: ITT Population included all participants who were randomized and had post-randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 281 | 425
months | 9.6 [8.67 to 11.99] | 17.8 [15.67 to 20.63]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.655, 95% CI 2-sided [0.537 to 0.799]; P-value comparing TTP between treatment groups was based on log-rank test stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR). Hazard ratio was based on an unadjusted Cox's proportional hazard regression model stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR), comparing the hazard rate of ixazomib arm over the hazard rate of placebo arm. A less than 1 hazard ratio was to be considered statistically significant

5. Secondary Outcome: Progression Free Survival 2 (PFS2)
Description: PFS2 is defined as the time from the date of randomization to objective PD on next-line treatment using IMWG criteria, or death due to any cause, whichever occurred first.
Time Frame: From the date of randomization to every 12 weeks until second PD or death (up to 88 months)
Population: ITT Population included all participants who were randomized and had post-randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 281 | 425
months | 50.3 [40.05 to 62.46] | 51.3 [44.91 to 63.41]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib; Test type: Superiority; p = 0.893, Log Rank; Hazard Ratio (HR) = 0.984, 95% CI 2-sided [0.777 to 1.246]; P-value comparing PFS2 between treatment groups was based on log-rank test stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR). Hazard ratio was based on an unadjusted Cox's proportional hazard regression model stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR), comparing the hazard rate of ixazomib arm over the hazard rate of placebo arm. A less than 1 hazard ratio was to be considered statistically significant

6. Secondary Outcome: Time to Next Line Therapy (TTNT)
Description: TTNT is defined as the time from the date of randomization to the date of the first dose of next-line antineoplastic therapy.
Time Frame: From randomization until PD or death (up to 52 months)
Population: ITT Population included all participants who were randomized and had post-randomization data.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 281 | 425
months | 16.1 [13.54 to 19.35] | 22.1 [19.55 to 25.89]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib; Test type: Superiority; p = 0.018, Log Rank; Hazard Ratio (HR) = 0.777, 95% CI 2-sided [0.631 to 0.957]; P-value comparing TTNT between treatment groups was based on log-rank test stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR). Hazard ratio was based on an unadjusted Cox's proportional hazard regression model stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR), comparing the hazard rate of ixazomib arm over the hazard rate of placebo arm. A less than 1 hazard ratio was to be considered statistically significant

7. Secondary Outcome: Time to End of the Next-line of Therapy After Study Treatment
Description: Time to end of the next line of therapy is defined as the time from the date of randomization to the date of last dose of the next line of antineoplastic therapy following study treatment.
Time Frame: From randomization until PD or death (up to 52 months)
Population: ITT Population included all participants who were randomized and had post-randomization data. Overall number analyzed is the number of participants with data available for analyses.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 164 | 215
months | 25.6 [22.70 to 28.48] | 23.1 [20.93 to 26.05]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib; Test type: Superiority; p = 0.462, Log Rank; Hazard Ratio (HR) = 1.111, 95% CI 2-sided [0.839 to 1.470]; P-value comparing Time to End of Next Line Therapy between treatment groups was based on log-rank test stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR). Hazard ratio was based on an unadjusted Cox's proportional hazard regression model stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR), comparing the hazard rate of ixazomib arm over the hazard rate of placebo arm. A less than 1 hazard ratio was to be considered statistically significant

8. Secondary Outcome: Duration of Next-line Therapy
Description: Duration of next-line therapy is defined as the time from the date of the first dose of the next line of antineoplastic therapy coming after study treatment to the date of the last dose.
Time Frame: From randomization until PD or death (up to 52 months)
Population: as for outcome 7
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 164 | 215
months | 14.0 [10.41 to 16.82] | 8.7 [7.85 to 10.87]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib; Test type: Superiority; Hazard Ratio (HR) = 1.293, 95% CI 2-sided [0.968 to 1.727]; Hazard ratio was based on an unadjusted Cox's proportional hazard regression model stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR), comparing the hazard rate of ixazomib arm over the hazard rate of placebo arm. A less than 1 hazard ratio was to be considered statistically significant

9. Secondary Outcome: Percentage of Participants Who Develop a New Primary Malignancy
Time Frame: From randomization until PD or death (up to 52 months)
Population: Safety Population included all participants who received at least 1 dose of ixazomib or placebo. Three placebo participants who erroneously received a single dose of ixazomib were included in the ixazomib arm of the safety population. The percentages are rounded off to the single nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 276 | 426
percentage of participants | 6.2 | 5.2

10. Secondary Outcome: Percentage of Participants With Conversion From Minimal Residual Disease (MRD) Positive to MRD Negative
Description: Bone marrow aspirates and blood samples were sent to a central laboratory and were assessed for MRD using flow cytometry. MRD negativity was defined as absence of MRD and MRD positivity was defined as presence of MRD. MRD was assessed by 8-color flow cytometry with the IMWG recommended sensitivity of 10^-5.
Time Frame: Up to 52 months
Population: ITT Population included all participants who were randomized and had post-randomization data. Overall number analyzed is the number of participants with data available for analyses. The percentages are rounded off to the nearest single decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 125 | 169
percentage of participants | 3 | 6

11. Secondary Outcome: Correlation of MRD Status With PFS and OS
Description: PFS is defined as the time from the date of randomization to the date of first documentation of PD or death from any cause, as evaluated by an IRC according to IMWG criteria, or death due to any cause, whichever occurred first, assessed for up to 52 months in this outcome measure. OS was measured as the time from the date of randomization to the date of death, assessed for up to 52 months in this outcome measure. Participants with various types of known MRD status were pooled together for analysis of overall survival in this outcome measure.
Time Frame: From randomization up to 52 months
Population: ITT Population included all participants who were randomized and had post-randomization data. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for the specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 151 | 213
months
  PFS for Participants with Known MRD+ at Study Entry: number analyzed (Participants) | 125 | 169
  PFS for Participants with Known MRD+ at Study Entry | 9.3 [7.75 to 11.99] | 16.9 [13.47 to 21.29]
  PFS for Participants with Known MRD- at Study Entry: number analyzed (Participants) | 26 | 44
  PFS for Participants with Known MRD- at Study Entry | NA [23.69 to NA] — Median and upper limit of confidence interval (CI) were not estimable due to censoring. | 40.5 [26.94 to NA] — Upper limit of CI was not estimable due to censoring.
  OS for Participants with Known MRD Status (MRD- Status, MRD+ Status) at Study Entry | NA [NA to NA] — Median, upper, and lower limit of CI were not estimable due to censoring. | NA [NA to NA] — Median, upper, and lower limit of CI were not estimable due to censoring.
Statistical Analysis 1: Comparison: Placebo vs Ixazomib; PFS for Participants with Known MRD+ at Study Entry; Test type: Superiority; p = 0.001, Log Rank; Hazard Ratio (HR) = 0.582, 95% CI 2-sided [0.425 to 0.796]; P-value comparing PFS between treatment groups was based on log-rank test stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR). Hazard ratio was based on an unadjusted Cox's proportional hazard regression model stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR), comparing the hazard rate of ixazomib arm over the hazard rate of placebo arm. A less than 1 hazard ratio was to be considered statistically significant
Statistical Analysis 2: Comparison: Placebo vs Ixazomib; PFS for Participants with Known MRD- at Study Entry; Test type: Superiority; p = 0.398, Log Rank; Hazard Ratio (HR) = 1.537, 95% CI 2-sided [0.563 to 4.194]; [other analysis details as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Ixazomib; OS for Participants with Known MRD Status (MRD- Status, MRD+ Status) at Study Entry; Test type: Superiority; p = 0.012, Log Rank; Hazard Ratio (HR) = 10.173, 95% CI 2-sided [1.194 to 86.649]; P-value comparing OS between treatment groups was based on log-rank test stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR). Hazard ratio was based on an unadjusted Cox's proportional hazard regression model stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), age (<75 vs >=75 years) at randomization, and best response to initial therapy (CR or VGPR vs PR), comparing the hazard rate of ixazomib arm over the hazard rate of placebo arm. A less than 1 hazard ratio was to be considered statistically significant

12. Secondary Outcome: OS in a High-risk Population
Description: High-risk population included but not be limited to participants carrying cytogenetic deletion (del)17, translocation [t](4;14), t(14;16). OS was measured as the time from the date of randomization to the date of death.
Time Frame: From the date of randomization and every 12 weeks after PD on next-line therapy until death (up to 88 months)
Population: ITT Population included all participants who were randomized and had post-randomization data. Overall number of participants analyzed is the number of participants present in the high-risk group.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 48 | 74
months | 48.3 [29.70 to 74.48] | 37.3 [26.05 to 47.44]

13. Secondary Outcome: PFS in a High-risk Population
Description: High-risk population included but not be limited to participants carrying del17, t(4;14), t(14;16). PFS was defined as the time from the date of randomization to the date of first documentation of PD or death from any cause.
Time Frame: From randomization until PD or death (up to 52 months)
Population: as for outcome 12
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 48 | 74
months | 9.6 [5.62 to 13.90] | 10.1 [6.01 to 17.02]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib; Test type: Superiority; p = 0.963, Log Rank; Hazard Ratio (HR) = 1.011, 95% CI 2-sided [0.631 to 1.621]; [other analysis details as in outcome 11, analysis 1]

14. Secondary Outcome: Change From Baseline in Eastern Cooperative Oncology Group (ECOG) Performance Status
Description: ECOG performance status assesses a participant's performance status on a 6-point scale ranging from 0=fully active/able to carry on all pre-disease activities without restriction; 1=restricted in physically strenuous activity, ambulatory/able to carry out light or sedentary work; 2=ambulatory (>50% of waking hours), capable of all self-care, unable to carry out any work activities; 3=capable of only limited self-care, confined to bed/chair >50% of waking hours; 4=completely disabled, cannot carry on any self-care, totally confined to bed/chair; 5=dead. Lower grades indicate improvement.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, and 26, progression free survival follow-up (PFSFU)- Visit 37 and progressive disease follow-up (PDFU)- Visit 26 (cycle length=28 days)
Population: Safety Population included all participants who received at least 1 dose of ixazomib or placebo. Three placebo participants who erroneously received a single dose of ixazomib were included in the ixazomib arm of the safety population. Overall number of participants analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for the specified category.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 271 | 415
score on a scale
  Cycle 2 Day 1 | -0.0 (0.36) | -0.0 (0.42)
  Cycle 3 Day 1: number analyzed (Participants) | 263 | 396
  Cycle 3 Day 1 | -0.0 (0.36) | -0.0 (0.42)
  Cycle 4 Day 1: number analyzed (Participants) | 251 | 379
  Cycle 4 Day 1 | -0.0 (0.39) | -0.1 (0.42)
  Cycle 5 Day 1: number analyzed (Participants) | 235 | 355
  Cycle 5 Day 1 | -0.0 (0.44) | -0.0 (0.44)
  Cycle 6 Day 1: number analyzed (Participants) | 219 | 332
  Cycle 6 Day 1 | -0.0 (0.46) | -0.0 (0.43)
  Cycle 7 Day 1: number analyzed (Participants) | 204 | 305
  Cycle 7 Day 1 | -0.0 (0.49) | -0.0 (0.42)
  Cycle 8 Day 1: number analyzed (Participants) | 188 | 287
  Cycle 8 Day 1 | -0.1 (0.48) | -0.0 (0.42)
  Cycle 9 Day 1: number analyzed (Participants) | 175 | 279
  Cycle 9 Day 1 | -0.1 (0.47) | -0.0 (0.45)
  Cycle 10 Day 1: number analyzed (Participants) | 163 | 261
  Cycle 10 Day 1 | -0.1 (0.52) | -0.0 (0.47)
  Cycle 11 Day 1: number analyzed (Participants) | 151 | 246
  Cycle 11 Day 1 | -0.1 (0.51) | -0.0 (0.43)
  Cycle 12 Day 1: number analyzed (Participants) | 142 | 235
  Cycle 12 Day 1 | -0.1 (0.56) | -0.0 (0.43)
  Cycle 13 Day 1: number analyzed (Participants) | 129 | 219
  Cycle 13 Day 1 | -0.0 (0.54) | -0.0 (0.46)
  Cycle 14 Day 1: number analyzed (Participants) | 115 | 204
  Cycle 14 Day 1 | 0.0 (0.53) | -0.0 (0.44)
  Cycle 15 Day 1: number analyzed (Participants) | 104 | 185
  Cycle 15 Day 1 | -0.0 (0.53) | -0.0 (0.49)
  Cycle 16 Day 1: number analyzed (Participants) | 96 | 177
  Cycle 16 Day 1 | -0.0 (0.51) | -0.0 (0.49)
  Cycle 17 Day 1: number analyzed (Participants) | 84 | 164
  Cycle 17 Day 1 | -0.0 (0.54) | -0.0 (0.50)
  Cycle 18 Day 1: number analyzed (Participants) | 74 | 159
  Cycle 18 Day 1 | 0.0 (0.51) | -0.0 (0.51)
  Cycle 19 Day 1: number analyzed (Participants) | 65 | 148
  Cycle 19 Day 1 | 0.0 (0.47) | -0.0 (0.49)
  Cycle 20 Day 1: number analyzed (Participants) | 57 | 133
  Cycle 20 Day 1 | 0.0 (0.46) | -0.0 (0.49)
  Cycle 21 Day 1: number analyzed (Participants) | 52 | 122
  Cycle 21 Day 1 | 0.0 (0.48) | -0.0 (0.52)
  Cycle 22 Day 1: number analyzed (Participants) | 51 | 111
  Cycle 22 Day 1 | 0.1 (0.51) | -0.0 (0.52)
  Cycle 23 Day 1: number analyzed (Participants) | 42 | 101
  Cycle 23 Day 1 | 0.0 (0.44) | -0.0 (0.48)
  Cycle 24 Day 1: number analyzed (Participants) | 41 | 91
  Cycle 24 Day 1 | 0.1 (0.54) | -0.0 (0.47)
  Cycle 25 Day 1: number analyzed (Participants) | 35 | 79
  Cycle 25 Day 1 | 0.0 (0.42) | -0.0 (0.47)
  Cycle 26 Day 1: number analyzed (Participants) | 28 | 68
  Cycle 26 Day 1 | 0.0 (0.47) | -0.0 (0.47)
  PFSFU- Visit 37: number analyzed (Participants) | 0 | 1
  PFSFU- Visit 37 |  | 1.0 (NA) — Standard deviation was not estimable for a single participant.
  PDFU- Visit 26: number analyzed (Participants) | 0 | 1
  PDFU- Visit 26 |  | 1.0 (NA) — Standard deviation was not estimable for a single participant.

15. Secondary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (e.g., a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. TEAEs were defined as events that occurred after administration of the first dose of ixazomib or placebo through 30 days after the last dose of ixazomib or placebo. A SAE means any untoward medical occurrence that resulted in death, was life-threatening, required in-patient hospitalization or prolongation of existing hospitalization, resulted in persistent or significant disability/incapacity, was a congenital anomaly/birth defect or was considered medically significant.
Time Frame: First dose of study drug through 30 days after last dose of study drug (up to 88 months)
Population: Safety Population included all participants who received at least 1 dose of ixazomib or placebo. Three placebo participants who erroneously received a single dose of ixazomib were included in the ixazomib arm of the safety population. The percentages were rounded off to the nearest single decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 276 | 426
percentage of participants
  SAE | 17 | 24
  TEAE | 82 | 92

16. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) as Measured by the Global Health Status (GHS)
Description: The EORTC QLQ-C30 is a questionnaire to assess the overall quality of life of cancer patients. The change from baseline in GHS (EORTC QLQ-C30) score is presented. Participant responses to the question "How would you rate your overall health during the past week?" are scored on a 7-point scale (1=very poor to 7=excellent). Using linear transformation, raw scores are standardized, so that scores range from 0 to 100. A higher score indicates a better overall GHS.
Time Frame: Baseline, Cycles 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, and 26 (cycle length=28 days)
Population: ITT Population included all participants who were randomized and had post-randomization data. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analyses for the specified time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 257 | 391
score on a scale
  Cycle 2 | 1.7 (16.63) | -0.1 (16.77)
  Cycle 3: number analyzed (Participants) | 257 | 375
  Cycle 3 | 2.1 (15.74) | -1.2 (17.14)
  Cycle 4: number analyzed (Participants) | 245 | 360
  Cycle 4 | 1.5 (16.80) | -0.6 (16.53)
  Cycle 5: number analyzed (Participants) | 227 | 340
  Cycle 5 | 1.8 (15.79) | 0.6 (16.33)
  Cycle 6: number analyzed (Participants) | 213 | 307
  Cycle 6 | 1.0 (18.33) | -1.5 (16.56)
  Cycle 7: number analyzed (Participants) | 202 | 292
  Cycle 7 | 3.1 (16.32) | -0.7 (17.28)
  Cycle 8: number analyzed (Participants) | 186 | 273
  Cycle 8 | 0.9 (18.07) | -0.4 (17.44)
  Cycle 9: number analyzed (Participants) | 173 | 258
  Cycle 9 | 1.4 (16.67) | 0.1 (16.57)
  Cycle 10: number analyzed (Participants) | 163 | 245
  Cycle 10 | 2.0 (16.38) | -1.6 (17.82)
  Cycle 11: number analyzed (Participants) | 152 | 233
  Cycle 11 | 3.9 (17.37) | 0.2 (17.75)
  Cycle 12: number analyzed (Participants) | 143 | 228
  Cycle 12 | 3.9 (14.53) | 0.3 (16.26)
  Cycle 13: number analyzed (Participants) | 132 | 218
  Cycle 13 | 4.2 (16.13) | -0.5 (16.85)
  Cycle 14: number analyzed (Participants) | 126 | 204
  Cycle 14 | 3.1 (16.99) | -1.1 (17.45)
  Cycle 15: number analyzed (Participants) | 115 | 194
  Cycle 15 | 2.2 (16.74) | -0.7 (17.65)
  Cycle 16: number analyzed (Participants) | 104 | 184
  Cycle 16 | 2.5 (15.57) | 0.5 (17.03)
  Cycle 17: number analyzed (Participants) | 100 | 182
  Cycle 17 | 2.4 (15.09) | -0.2 (18.09)
  Cycle 18: number analyzed (Participants) | 91 | 182
  Cycle 18 | 0.5 (18.40) | 1.7 (16.87)
  Cycle 19: number analyzed (Participants) | 82 | 172
  Cycle 19 | 1.6 (18.07) | 1.1 (17.24)
  Cycle 20: number analyzed (Participants) | 74 | 161
  Cycle 20 | 1.1 (17.95) | 0.4 (16.13)
  Cycle 21: number analyzed (Participants) | 72 | 153
  Cycle 21 | 1.5 (16.39) | 1.3 (16.19)
  Cycle 22: number analyzed (Participants) | 72 | 147
  Cycle 22 | 1.6 (15.55) | 1.0 (17.13)
  Cycle 23: number analyzed (Participants) | 68 | 137
  Cycle 23 | 2.1 (19.01) | 0.9 (16.96)
  Cycle 24: number analyzed (Participants) | 64 | 132
  Cycle 24 | -0.3 (20.46) | 2.3 (15.65)
  Cycle 25: number analyzed (Participants) | 56 | 125
  Cycle 25 | 0.0 (18.80) | 0.3 (17.52)
  Cycle 26: number analyzed (Participants) | 47 | 106
  Cycle 26 | 2.8 (17.49) | 0.9 (17.26)

17. Secondary Outcome: Correlation Between Frailty Status and PFS and OS
Description: Participant's frailty status is classified as fit, unfit or frail on the bases of 4 components: age, the Charlson comorbidity scoring system without age weighting, the Katz index of independence in activities of daily living, and the Lawton instrumental activities of daily living scale. The sum of the 4 frailty scores equals the total frailty score. A total frailty score of 0 corresponds to a frailty status of fit; a total score of 1, to unfit; and a total score of 2 or more, to frail. PFS is defined as the time from the date of randomization to the date of first documentation of PD or death from any cause, as evaluated by an IRC according to IMWG criteria, or death due to any cause, whichever occurs first, assessed for up to 52 months in this outcome measure. OS will be measured as the time from the date of randomization to the date of death, assessed for up to 52 months in this outcome measure.
Time Frame: From randomization up to 52 months
Population: ITT Population included all participants who were randomized and had post-randomization data. Overall number analyzed is the number of participants with data available for analyses. Number analyzed is the number of participants with data available for analysis for the specified category.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 112 | 172
months
  PFS Based on Frailty Status of Fit | 8.5 [7.39 to 10.41] | 18.6 [12.75 to 25.63]
  PFS Based on Frailty Status of Unfit: number analyzed (Participants) | 98 | 147
  PFS Based on Frailty Status of Unfit | 10.6 [7.39 to 14.23] | 17.6 [13.17 to 21.78]
  PFS Based on Frailty Status of Frail: number analyzed (Participants) | 68 | 102
  PFS Based on Frailty Status of Frail | 11.1 [8.44 to 15.67] | 15.4 [11.10 to 23.75]
  OS Based on Frailty Status of Fit | NA [NA to NA] — Median, upper, and lower limit of CI were not estimable due to censoring. | NA [NA to NA] — Median, upper, and lower limit of CI were not estimable due to censoring.
  OS Based on Frailty Status of Unfit: number analyzed (Participants) | 98 | 147
  OS Based on Frailty Status of Unfit | NA [NA to NA] — Median, upper, and lower limit of CI were not estimable due to censoring. | NA [39.59 to NA] — Median and lower limit of CI were not estimable due to censoring.
  OS Based on Frailty Status of Frail: number analyzed (Participants) | 68 | 102
  OS Based on Frailty Status of Frail | 42.5 [29.93 to NA] — Upper limit of CI was not estimable due to censoring. | 46.5 [34.30 to 46.52]
Statistical Analysis 1: Comparison: Placebo vs Ixazomib; PFS Based on Frailty Status of Fit; Test type: Superiority; p < 0.001, Log Rank; Hazard Ratio (HR) = 0.530, 95% CI 2-sided [0.387 to 0.727]; P-value comparing PFS between treatment groups was based on Log-rank test stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), and age (<75 vs >=75 years) at randomization. Hazard ratio was based on an unadjusted Cox's proportional hazard regression model stratified by initial therapy (proteasome inhibitor-containing or not), ISS stage before initial therapy (stage I or II vs stage III), and age (<75 vs >=75 years) at randomization, comparing the hazard rate of ixazomib arm over the hazard rate of placebo arm. A less than 1 hazard ratio was to be considered statistically significant
Statistical Analysis 2: Comparison: Placebo vs Ixazomib; PFS Based on Frailty Status of Unfit; Test type: Superiority; p = 0.098, Log Rank; Hazard Ratio (HR) = 0.746, 95% CI 2-sided [0.526 to 1.058]; [other analysis details as in outcome 17, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Ixazomib; PFS Based on Frailty Status of Frail; Test type: Superiority; p = 0.147, Log Rank; Hazard Ratio (HR) = 0.733, 95% CI 2-sided [0.481 to 1.117]; [other analysis details as in outcome 17, analysis 1]
Statistical Analysis 4: Comparison: Placebo vs Ixazomib; OS Based on Frailty Status of Fit; Test type: Superiority; p = 0.714, Log Rank; Hazard Ratio (HR) = 0.897, 95% CI 2-sided [0.502 to 1.602]; [other analysis details as in outcome 11, analysis 3]
Statistical Analysis 5: Comparison: Placebo vs Ixazomib; OS Based on Frailty Status of Unfit; Test type: Superiority; p = 0.124, Log Rank; Hazard Ratio (HR) = 1.750, 95% CI 2-sided [0.850 to 3.601]; [other analysis details as in outcome 11, analysis 3]
Statistical Analysis 6: Comparison: Placebo vs Ixazomib; OS Based on Frailty Status of Frail; Test type: Superiority; p = 0.630, Log Rank; Hazard Ratio (HR) = 0.854, 95% CI 2-sided [0.448 to 1.627]; [other analysis details as in outcome 11, analysis 3]

18. Secondary Outcome: Pharmacokinetic Parameter: Plasma Concentration of Ixazomib
Description: Plasma concentrations of the complete hydrolysis product of ixazomib citrate (ixazomib) were measured using a validated liquid chromatography-tandem mass spectrometry (LC/MS/MS) assay.
Time Frame: Cycle 1 (1 and 4 hours post-dose Day 1, Days 8 and 15 pre-dose); Cycle 2 and 5 (Days 1 and 8 pre-dose) and Cycles 3, 4, 6 to 10 (Day 1 pre-dose) (cycle length=28 days)
Population: Pharmacokinetic Analysis Population included all participants with at least one pharmacokinetic (PK) sample that was collected and analyzed. Number analyzed is the number of participants with data available for analysis at the specified time point.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Ixazomib
Number analyzed (Participants) | 423
nanogram per milliliter (ng/mL)
  Cycle 1 Day 1 - 1 Hour Post-dose: number analyzed (Participants) | 413
  Cycle 1 Day 1 - 1 Hour Post-dose | 19.353 (89.2568)
  Cycle 1 Day 1 - 4 Hours Post-dose: number analyzed (Participants) | 403
  Cycle 1 Day 1 - 4 Hours Post-dose | 12.698 (67.8350)
  Cycle 1 Day 8 - Pre-dose: number analyzed (Participants) | 409
  Cycle 1 Day 8 - Pre-dose | 1.683 (162.3947)
  Cycle 1 Day 15 - Pre-dose: number analyzed (Participants) | 411
  Cycle 1 Day 15 - Pre-dose | 2.828 (86.7699)
  Cycle 2 Day 1 - Pre-dose: number analyzed (Participants) | 410
  Cycle 2 Day 1 - Pre-dose | 1.958 (170.8938)
  Cycle 2 Day 8 - Pre-dose: number analyzed (Participants) | 394
  Cycle 2 Day 8 - Pre-dose | 3.217 (188.6379)
  Cycle 3 Day 1 - Pre-dose: number analyzed (Participants) | 391
  Cycle 3 Day 1 - Pre-dose | 2.252 (56.2869)
  Cycle 4 Day 1 - Pre-dose: number analyzed (Participants) | 372
  Cycle 4 Day 1 - Pre-dose | 2.363 (52.9781)
  Cycle 5 Day 1 - Pre-dose: number analyzed (Participants) | 348
  Cycle 5 Day 1 - Pre-dose | 2.328 (53.0909)
  Cycle 5 Day 8 - Pre-dose: number analyzed (Participants) | 257
  Cycle 5 Day 8 - Pre-dose | 4.547 (224.4312)
  Cycle 6 Day 1 - Pre-dose: number analyzed (Participants) | 320
  Cycle 6 Day 1 - Pre-dose | 2.503 (52.9349)
  Cycle 7 Day 1 - Pre-dose: number analyzed (Participants) | 298
  Cycle 7 Day 1 - Pre-dose | 2.585 (57.9514)
  Cycle 8 Day 1 - Pre-dose: number analyzed (Participants) | 281
  Cycle 8 Day 1 - Pre-dose | 2.606 (58.5109)
  Cycle 9 Day 1 - Pre-dose: number analyzed (Participants) | 269
  Cycle 9 Day 1 - Pre-dose | 2.566 (58.1094)
  Cycle 10 Day 1 - Pre-dose: number analyzed (Participants) | 250
  Cycle 10 Day 1 - Pre-dose | 2.686 (50.2494)

19. Secondary Outcome: Time to Resolution of Peripheral Neuropathy (PN) Events
Description: PN is defined as the event in the high-level term of peripheral neuropathies not elsewhere classified (NEC) according to the medical dictionary for regulatory activities (MedDRA). A PN event was considered as resolved if its final outcome was resolved with no subsequent PN event of the same preferred term occurring on the resolution date or the day before and after. Time to resolution was defined as the time from the initial onset date (inclusive) to the resolution date for resolved events.
Time Frame: Up to 52 months
Population: Safety Population included all participants who received at least 1 dose of ixazomib or placebo. Overall number of participants analyzed are the number of participants with events.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 30 | 83
days | 196.0 [43.0 to 331.0] | 451.0 [98.0 to NA] — Upper limit of CI was not estimable due to censoring.

20. Secondary Outcome: Time to Improvement of PN Events
Description: PN is defined as the event in the high-level term of peripheral neuropathies NEC according to the MedDRA. A PN event was considered as resolved if its final outcome was resolved with no subsequent PN event of the same preferred term occurring on the improvement date or the day before and after. Time to improvement was defined as the time from the initial onset date (inclusive) to the improvement of event.
Time Frame: Up to 52 months
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Placebo | Ixazomib
Number analyzed (Participants) | 30 | 83
days | 81.0 [15.0 to 280.0] | 64.0 [29.0 to 393.0]

ADVERSE EVENTS:
Time Frame: First dose of study drug through 30 days after last dose of study drug (up to 88 months)
Description: All-cause mortality= ITT Population included all participants who were randomized and had post-randomization data. Serious and Other Adverse Events: Safety population included all participants who received at least 1 dose of ixazomib or placebo. Three participants assigned to placebo arm each received a single 3 mg dose of ixazomib. These participants were excluded from the placebo arm and included in the ixazomib arm in the safety population.
Arm/Group | Placebo | Ixazomib
All-Cause Mortality (participants affected / at risk) | 115/281 | 184/425
Serious Adverse Events (participants affected / at risk) | 48/276 | 101/426
Other Adverse Events (participants affected / at risk) | 188/276 | 340/426
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=276) | Ixazomib (N=426)
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 5
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 3 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Atrial tachycardia (Cardiac disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 3
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Bronchiolitis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cardiac arrest (Cardiac disorders) | 0 | 1
Cardiac failure (Cardiac disorders) | 0 | 1
Cardiac failure acute (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Chest pain (General disorders) | 0 | 1
Chilaiditi's syndrome (Gastrointestinal disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Chronic kidney disease (Renal and urinary disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Coronary artery disease (Cardiac disorders) | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Gastric disorder (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis radiation (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastrointestinal motility disorder (Gastrointestinal disorders) | 0 | 1
General physical health deterioration (General disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 0 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertensive emergency (Vascular disorders) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 0 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 1
Jugular vein thrombosis (Vascular disorders) | 0 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 5
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Melaena (Gastrointestinal disorders) | 0 | 1
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Monoparesis (Nervous system disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 2 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 2
Non-small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Paraneoplastic pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Partial seizures (Nervous system disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 2 | 3
Pelvic fracture (Injury, poisoning and procedural complications) | 2 | 0
Pericardial effusion (Cardiac disorders) | 0 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 5
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 16
Pneumonia viral (Infections and infestations) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Pyrexia (General disorders) | 1 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1
Rectal prolapse (Gastrointestinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Rhinovirus infection (Infections and infestations) | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Sepsis (Infections and infestations) | 0 | 3
Septic shock (Infections and infestations) | 1 | 4
Soft tissue injury (Injury, poisoning and procedural complications) | 0 | 1
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Subcapsular renal haematoma (Renal and urinary disorders) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 0
Sudden death (General disorders) | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Transient ischaemic attack (Nervous system disorders) | 1 | 2
Transitional cell cancer of the renal pelvis and ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Trismus (Musculoskeletal and connective tissue disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 6
Uveitis (Eye disorders) | 1 | 0
Varicella (Infections and infestations) | 0 | 1
Vomiting (Gastrointestinal disorders) | 2 | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=276) | Ixazomib (N=426)
Anaemia (Blood and lymphatic system disorders) | 19 | 31
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 61
Asthenia (General disorders) | 17 | 25
Back pain (Musculoskeletal and connective tissue disorders) | 33 | 62
Constipation (Gastrointestinal disorders) | 21 | 36
Cough (Respiratory, thoracic and mediastinal disorders) | 19 | 31
Decreased appetite (Metabolism and nutrition disorders) | 13 | 36
Diarrhoea (Gastrointestinal disorders) | 35 | 102
Dizziness (Nervous system disorders) | 16 | 27
Dyspepsia (Gastrointestinal disorders) | 7 | 24
Fatigue (General disorders) | 28 | 49
Headache (Nervous system disorders) | 11 | 23
Hypertension (Vascular disorders) | 16 | 26
Insomnia (Psychiatric disorders) | 12 | 26
Myalgia (Musculoskeletal and connective tissue disorders) | 8 | 22
Nasopharyngitis (Infections and infestations) | 18 | 36
Nausea (Gastrointestinal disorders) | 23 | 119
Oedema peripheral (General disorders) | 16 | 37
Pain in extremity (Musculoskeletal and connective tissue disorders) | 13 | 25
Peripheral sensory neuropathy (Nervous system disorders) | 25 | 66
Pruritus (Skin and subcutaneous tissue disorders) | 12 | 24
Pyrexia (General disorders) | 13 | 44
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 36
Upper respiratory tract infection (Infections and infestations) | 32 | 69
Vomiting (Gastrointestinal disorders) | 11 | 102

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT02312258/Prot_002.pdf
  • Statistical Analysis Plan (2019-09-20): https://cdn.clinicaltrials.gov/large-docs/58/NCT02312258/SAP_000.pdf